CLINICAL TRIAL: NCT01543334
Title: Antibiotic Concentrations Among Critically Ill Patients
Acronym: DALI
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2011/JYL-03; 2011-A01339-32 (Other: ANSM)
Record Dates: First submitted 2012-02-20; First posted 2012-03-02 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2015-03

CONDITIONS: Administration of Antibiotics in Intensive Care Units
Keywords: intensive care; antibiotic levels in blood samples
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients: Patients with a vein or artery catheter and who are being administered antibiotics. The latter can be of the following: Amoxicillin-clavulanic acid, ampicillin, piperacillin-tazobactam, penicillin G, flucloxacillin, dicloxacillin, cloxacillin, cefazolin, ceftazidime, ceftriaxone, cefepime, meropenem, imipenem, doripenem, ertapenem; Vancomycin, teicoplanin. (see inclusion/exclusion criteria).
  Interventions: Biological: Blood sampling

INTERVENTIONS:
Biological: Blood sampling — Blood samples will be harvested in one sequence at any time during the week set for the study. In patients receiving multiple antibiotics, multiple samples can be made (without exceeding the study of three antibiotics, ie a maximum of 6 tubes per patient). Two 3-ml tubes of blood will be collected for beta-lactams and glycopeptides (Sample A taken at half the time of the dosing interval and sample B at 30 minutes before the next dose). When patients receive continuous antibiotic treatment, both samples must be made at least 6 hours apart.

SUMMARY:
The primary objective of the DALI study is to compare antibiotic concentrations in patient blood samples with bacteriological objectives associated with maximum bactericidal activity. The antibiotics studied are certain lactams and glycopeptides.

ELIGIBILITY:
Inclusion Criteria:

* The patient (or his/her "trusted representative") must have given his/her informed and signed consent
* Antibiotic treatment is administered with beta-lactams or glycopeptides administered continuously or intermittently (Can be of the following: Amoxicillin-clavulanic acid, ampicillin, piperacillin-tazobactam, penicillin G, flucloxacillin, dicloxacillin, cloxacillin, cefazolin, ceftazidime, ceftriaxone, cefepime, meropenem, imipenem, doripenem, ertapenem; Vancomycin, teicoplanin).
* A vein or artery catheter is established to facilitate blood sampling (arterial catheter is preferred)

Exclusion Criteria:

* None of the above-mentioned antibiotics are administered
* Impossible to establish venous or arterial catheter
* Consent not given
* Patient is pregnant, parturient or breastfeeding
* The patient is under tutorship or curatorship
* The patient is participating in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive care patients with a vein or artery catheter and who are being administered antibiotics Can be of the following: Amoxicillin-clavulanic acid, ampicillin, piperacillin-tazobactam, penicillin G, flucloxacillin, dicloxacillin, cloxacillin, cefazolin, ceftazidime, ceftriaxone, cefepime, meropenem, imipenem, doripenem, ertapenem; Vancomycin, teicoplanin.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2012-03; Primary Completion 2012-04-01 (Actual); Study Completion 2012-04-01 (Actual)

PRIMARY OUTCOMES:
[antibiotics] in blood versus bactericidal activity | 1/2 antibiotic dose interval (expected maximum of 4 days; days 1 to 4)
  The primary endpoint for the DALI study is the comparison of antibiotic concentrations in patient blood samples with bacteriological objectives associated with maximum bactericidal activity. The antibiotics studied are certain lactams (endpoint pharmacokinetics 50 and 100% T> MIC) and glycopeptides (100% T> 4xCMI and report ASC0-24/CMI ≥ 350).
[antibiotics] in blood versus bactericidal activity | 30 minutes before second antibiotic dose (expected maximum of 7 days; days 1 to 7)
  The primary endpoint for the DALI study is the comparison of antibiotic concentrations in patient blood samples with bacteriological objectives associated with maximum bactericidal activity. The antibiotics studied are certain lactams (endpoint pharmacokinetics 50 and 100% T> MIC) and glycopeptides (100% T> 4xCMI and report ASC0-24/CMI ≥ 350).

SECONDARY OUTCOMES:
Apache II score | at time of blood sampling (day 1)
SOFA score | at time of blood sampling (day 1)
PIRO score | at time of blood sampling (day 1)
Diagnosis at admission | Admission to ICU (day 1)
Indication for antibiotic treatment | at time of blood sampling (day 1)
did the patient have a surgical procedure in the last 24 hours? | at time of blood sampling (day 1)
  yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Jean Yves Lefrant, MD PhD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (13):
- France (13):
  - CH du Pays d'Aix, Aix-en-Provence
  - CHU d'Amiens - Hôpital Nord, Amiens
  - CHU d'Angers - Hôtel-Dieu, Angers
  - CHU de Clermont Ferrand - Hôpital Estaing, Clermont-Ferrand
  - CHU de Grenoble - Hôpital A Michallon, Grenoble
  - APHM - Hôpital Nord, Marseille
  - CHU de Montpellier - Hôpital Saint-Eloi, Montpellier
  - CHU de Nice - Hôpital St-Roch, Nice
  - CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes
  - APHP - Hôpital Bichat - Claude Bernard, Paris
  - CHU de Bordeaux - Hôpital Haut-Lévêque, Pessac
  - CHU de Rennes - Hôpital PontChaillou, Rennes
  - CHRU de Strasbourg - Hôpital Civil, Strasbourg

REFERENCES:
- [Result] Roberts JA, Paul SK, Akova M, Bassetti M, De Waele JJ, Dimopoulos G, Kaukonen KM, Koulenti D, Martin C, Montravers P, Rello J, Rhodes A, Starr T, Wallis SC, Lipman J; DALI Study. DALI: defining antibiotic levels in intensive care unit patients: are current beta-lactam antibiotic doses sufficient for critically ill patients? Clin Infect Dis. 2014 Apr;58(8):1072-83. doi: 10.1093/cid/ciu027. Epub 2014 Jan 14. PMID 24429437